CLINICAL TRIAL: NCT03400345
Title: Human Upper Extremity Allotransplantation: Transplanted Patient Follow-Up Protocol
Brief Title: Human Upper Extremity Allotransplantation: F/U Protocol
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00068053
Record Dates: First submitted 2017-10-13; First posted 2018-01-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Amputation, Traumatic; Wounds and Injury; Hand Injuries
Keywords: Hand Transplant; composite tissue allograft (CTA); Vascularized Composite Allotransplantation (VCA); Amputation; Upper Limb; Immunosuppression
MeSH Terms: conditions — Amputation, Traumatic; Wounds and Injuries; Hand Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Upper extremity allotransplantation is a new procedure which is becoming more common in the United States. Ongoing data collection for research purposes is vital to the long-term assessment as to the safety of the procedure and accompanying immunosuppression protocol, as well as quantifying patient outcomes and changes in quality of life. For these reasons, The Johns Hopkins Hand/Arm Transplantation Team is interested in enrolling transplanted patients in a follow-up protocol to continue collecting informative data to further the field of vascularized composite allotransplantation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 5 or more years post-unilateral or bilateral upper limb transplantation.
* Completes the protocol informed consent form.
* Consents to sample collection and storage (biopsies).
* USA citizen or equivalent.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regime.

Exclusion Criteria:

* Candidate has not received an upper extremity allotransplant.
* Any reason the study team thinks would cause the participant to be noncompliant or would put the patient at unacceptable risk if enrolled.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women who have previously received unilateral or bilateral upper limb transplants.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2036-07-30 (Estimated); Study Completion 2036-07-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) for upper extremity transplant recipients via Functional Assessment with rehabilitation using Carroll Test | Change from baseline QOL at end of study (approximately 5 years post-enrollment (±90 days))
  Measures Grasp, Grip and Pinch Strength, Range of motion - Active & Passive. During rehabilitation sessions in clinic using activities resembling everyday tasks such as pouring water, opening/closing zippers and buttons, lifting blocks of different weight. Carroll test contains 33 questions and is scored from 0-3, 0- can perform no part of test, 1- performs test partially, 2-completes test, but takes abnormally long time or has great difficulty, and 3- performs tests normally.
QOL assessed for Hand Function by Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Change from baseline QOL at end of study (approximately 5 years post-enrollment (±90 days))
  The DASH Outcome Measure is scored in two components: the disability/symptom section (30 items, scored 1-5) and the optional high performance Sport/Music or Work section (4 items, scored 1-5). 1 indicating no difficulty and 5 indicating unable perform the function.
QOL assessed by Lawton Instrumental Activities of Daily Living (ADL/IADL) Questionnaire | Change from baseline QOL at end of study (approximately 5 years post-enrollment (±90 days))
  Questionnaire to asses Physical and instrumental activities for daily living. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning). The scale will vary along a range of levels of competence- without any help, with some help, or does he need someone for the activities.
Michigan Hand Outcomes Questionnaire | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  Monitor function, pain, work performance, and aesthetics of hand(s). Responses from 1-5, 1 being very good and 5 being very poor
Short Musculoskeletal Function Assessment (SMFA) | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  The SMFA consists of two sections: 34 questions covering the assessment of the patients function and 12 questions covering how bothered patients are by their symptoms. Each question is scored 1 for no problems/no difficulty/not bothered (depending on the question) to 5 for unable to do a task/symptoms all the time/being greatly bothered.
Brief Pain Inventory (Short Form) (BPISF) | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  BPISF assesses the severity of pain and its impact on functioning. It is scored from 0 to 10, 0 indicating no pain, does not interfere to 10 indicating pain as bad as you can imagine, completely interferes.
Quality of life assessed for Psychological Measures by Brief Symptom Inventory | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  Brief Symptom Inventory questionnaire evaluates psychological distress and psychiatric disorders. It consists of 53-item self-report inventory in which participants rate the extent to which they have been bothered. 5-point rating scale, 0 indicating not at all bothered to 4 extremely bothered.
Psychological Measures by Satisfaction with Life Scale (SWLS) | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  SWLS is a measure of life satisfaction. Uses scale to rate from 1-7, Where 1 indicates Strongly disagree to 7 indicating strongly agree.
Psychological Measures assessed by Affect Balance Scale (ABS) | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  ABS is a 10-item questionnaire that assess positive and negative affect as indicators of life satisfaction and/or well-being. Score range from 0-4. 0 indicating the feeling never affected to 4, where the feeling is affected always.
Psychological Measures assessed by NEO Five-Factor Inventory (NEO-FFI) | Change from baseline to end of study (approximately 5 years post-enrollment (±90 days))
  NEO-FFI is used to examine personality traits. Questions consists of 60 items. Items are scored from Strongly disagree to Strongly agreed

SECONDARY OUTCOMES:
The efficacy of various immunosuppression regimens via ImmuKnow Assay/Cylex including immunomodulatory protocols (aka - Pittsburgh Protocol, Starzl Protocol), for maintenance of unilateral and bilateral upper extremity allotransplants. | Annually for 5 years post-enrollment (±90 days)
  For immune monitoring, to test cell mediated immunity. Value of ≤ 225 ng/mL indicates Low immune cell response, 226-524 ng/mL- Moderate Immune response, ≥525 ng/mL- High Immune cell Response.
Immunology- antibody testing by obtaining donor specific antibodies (DSA) by Luminex | Annually for 5 years (±90 days)
  For immune monitoring, to screen for donor specific antibodies.
Perform Skin Biopsy | Annually for 5 years (±90 days)
  To diagnose and assess acute rejection, Graft versus Host Disease and for surveillance of chronic rejection
Use CT Angiography | Annually for 5 years (±90 days)
  To delineate the outline and architecture of vasculature and blood flow patterns in the limb.
Magnetic Resonance (MR) Neurography | Annually for 5 years (±90 days)
  To help assess progression of nerve regeneration distal to the site of transplanted nerve coaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Shores, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Pooled patient data will be shared.

REFERENCES:
- [Background] Shores JT, Malek V, Lee WPA, Brandacher G. Outcomes after hand and upper extremity transplantation. J Mater Sci Mater Med. 2017 May;28(5):72. doi: 10.1007/s10856-017-5880-0. Epub 2017 Mar 30. PMID 28361279
- [Background] Shores JT, Brandacher G, Lee WPA. Hand and upper extremity transplantation: an update of outcomes in the worldwide experience. Plast Reconstr Surg. 2015 Feb;135(2):351e-360e. doi: 10.1097/PRS.0000000000000892. PMID 25401735
- [Background] Adler BL, Albayda J, Shores JT, Lee WPA, Brandacher G, Bingham CO 3rd. Erosive Rheumatoid Arthritis After Bilateral Hand Transplantation. Ann Intern Med. 2017 Aug 1;167(3):216-218. doi: 10.7326/L16-0588. Epub 2017 Jun 27. No abstract available. PMID 28654973
- See also: Human Upper Extremity Allotransplantation — https://www.hopkinsmedicine.org/transplant/programs/reconstructive-transplant/hand-arm-transplant